CLINICAL TRIAL: NCT00751270
Title: A Phase 1b Study of AdV-tk + Valacyclovir Gene Therapy in Combination With Standard Radiation Therapy for Malignant Gliomas
Brief Title: Phase 1b Study of AdV-tk + Valacyclovir Combined With Radiation Therapy for Malignant Gliomas
Acronym: BrTK01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrTK01
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: Immunotherapy; Gene therapy; Tumor Vaccine; Cytotoxicity; Radiation
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Arm A for unresectable malignant glioma was closed due to poor accrual.
  Interventions: Biological: AdV-tk; Drug: Valacyclovir
- B (Experimental): Arm B for resectable malignant glioma completed the Phase I accrual and long term follow up continues. A follow on study at dose level 3 was opened as a Phase 2a study (see BrTK02).
  Interventions: Biological: AdV-tk; Drug: Valacyclovir

INTERVENTIONS:
Biological: AdV-tk — Three different dosing levels of AdV-tk (3x10e10, 1x10e11, 3X10e11) were evaluated. A single injection of AdV-tk at the assigned dose level was administered, followed by 14 days of the oral prodrug valacyclovir. Patients then received standard of care radiation therapy and chemotherapy.
Drug: Valacyclovir — The oral prodrug valacyclovir was given beginning 1-3 days following the AdV-tk. Valacyclovir tablets were taken three times a day for a total of 14 days.

SUMMARY:
This phase I study evaluated a Gene Mediated Cytotoxic Immunotherapy approach for malignant gliomas, including glioblastoma multiforme and anaplastic astrocytoma. The purpose of this study was to assess the safety and feasibility of delivering an experimental approach called GliAtak which uses AdV-tk, an adenoviral vector containing the Herpes Simplex thymidine kinase gene, plus an oral anti-herpetic prodrug, valacyclovir, in combination with standard of care radiation.

DETAILED DESCRIPTION:
This study was designed to include patients with newly diagnosed unresectable (Arm A) and resectable (Arm B) malignant glioma. Three dose levels of AdV-tk were evaluated with a fixed dose level of valacyclovir prodrug. AdV-tk was delivered to tumor cells by stereotactic injection into the tumor at the time of biopsy (Arm A) or injection into the tumor bed following resection (Arm B). Oral valacyclovir began 1-3 days after the AdV-tk injection and continued for 14 days. Standard radiation therapy began 3-7 days following the AdV-tk injection to maximize synergy with radiation. Standard temozolomide could be administered after completion of valacyclovir.

ELIGIBILITY:
Inclusion Criteria:

* Presumed malignant glioma based on clinical and radiologic evaluation (pathologic confirmation of malignant glioma must be made at the time of stereotactic biopsy or resection prior to AdV-tk injection; if this is not possible, the injection will not be performed and the subject will no longer be eligible for the study).
* Tumor must be accessible for injection and must not be located in the brainstem, midbrain, contained within the ventricular system, or located in an infratentorial location.
* Patients must be planning to undergo standard radiation therapy.
* Patients must be 18 years of age or older.
* Performance status must be KPS > or equal to 70.
* Patients must have SGOT (AST) < 3x upper limit of normal.
* Patients must have serum creatinine < 2mg/dl and calculated creatinine clearance >10ml/min.
* Patients must have platelets > 100,000/mm3 and WBC > 3000/mm3.
* Patients of reproductive age must agree to use a medically accepted form of birth control while on the study.
* Patients must give study specific informed consent prior to enrollment.
* Patients must be able to tolerate MRI scan procedure

Exclusion Criteria:

* Prior or ongoing liver disease including known cirrhosis, hepatitis B or C infection but not to exclude patients with a distant history of resolved hepatitis A infection.
* Patients on immunosuppressive drugs (with exception of corticosteroid)
* Known HIV+ patients.
* Patients with acute infections (viral, bacterial or fungal infections requiring therapy).
* Pregnant or breast feeding patients. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy.
* Evidence of metastatic disease or other malignancy (except squamous or basal cell skin cancers).
* Prior radiation therapy to the brain or prior treatment for brain tumor (except prior biopsy or subtotal resection).
* Other serious co-morbid illness or compromised organ function.
* Patients may not receive temozolomide until valacyclovir completed and may not receive other investigational anti-tumor agents within 30 days prior to study entry or during active participation in the study (defined as from study entry until tumor progression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Through month 3 and long term follow up for late effects.

SECONDARY OUTCOMES:
Progression-free Survival | Clinical monitoring, laboratory and radiological imagining and pathological/histological assessments (if performed)
Overall Survival | 5 years
Functional Assessment of Cancer Therapy - Brain (FACT-Br) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: E. Antonio Chiocca, MD, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Dept Neurosurgery, Columbus, Ohio
  - The Methodist Hosptial, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chiocca EA, Aguilar LK, Bell SD, Kaur B, Hardcastle J, Cavaliere R, McGregor J, Lo S, Ray-Chaudhuri A, Chakravarti A, Grecula J, Newton H, Harris KS, Grossman RG, Trask TW, Baskin DS, Monterroso C, Manzanera AG, Aguilar-Cordova E, New PZ. Phase IB study of gene-mediated cytotoxic immunotherapy adjuvant to up-front surgery and intensive timing radiation for malignant glioma. J Clin Oncol. 2011 Sep 20;29(27):3611-9. doi: 10.1200/JCO.2011.35.5222. Epub 2011 Aug 15. PMID 21844505
- See also: Phase IB study of gene-mediated cytotoxic immunotherapy adjuvant to up-front surgery and intensive timing radiation for malignant glioma — http://www.ncbi.nlm.nih.gov/pubmed/21844505